CLINICAL TRIAL: NCT01429064
Title: Safety and Tolerability of ODM-201 in Patients With Castrate Resistant Prostate Cancer: Open, Non-randomised, Uncontrolled, Multicentre, Extension Study to Study 3104001
Brief Title: Safety and Tolerability of ODM-201 in Castrate Resistant Prostate Cancer; Extension Study to Study 3104001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3104002
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Results first posted 2016-12-22 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ODM-201 (Experimental)
  Interventions: Drug: ODM-201

INTERVENTIONS:
Drug: ODM-201 — ODM-201 administered orally daily

SUMMARY:
The purpose of this study is to evaluate safety and tolerability of ODM-201 in patients with castrate resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Successful completion of study protocol 3104001
* Response or stable disease in study 3104001 at week 12

Exclusion Criteria:

* New serious concurrent medical condition
* Not able to swallow the study drug

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karim Fizazi, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (17):
- United States (4):
  - The Urology Center of Colorado, Wheat Ridge, Colorado
  - Eastern CT Hematology and Oncology Associates, Norwich, Connecticut
  - Cleveland Clinic, Cleveland, Ohio
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
- Klinika onkologie a radioterapie LFUK a FN, Hradec Králové, Czechia
- East-Tallinn Central Hospital, Tallinn, Estonia
- Finland (5):
  - Helsinki University Central Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- France (2):
  - Saint Louis Hospital, Paris
  - Institut Gustave Roussy, Villejuif
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - Velindre Cancer Centre, Cardiff
  - Christie Hospital, Manchester
  - Churchill Hospital, Oxford

REFERENCES:
- [Derived] Shore ND, Tammela TL, Massard C, Bono P, Aspegren J, Mustonen M, Fizazi K. Safety and Antitumour Activity of ODM-201 (BAY-1841788) in Chemotherapy-naive and CYP17 Inhibitor-naive Patients: Follow-up from the ARADES and ARAFOR Trials. Eur Urol Focus. 2018 Jul;4(4):547-553. doi: 10.1016/j.euf.2017.01.015. Epub 2017 Feb 14. PMID 28753851
- [Derived] Fizazi K, Massard C, Bono P, Kataja V, James N, Tammela TL, Joensuu H, Aspegren J, Mustonen M. Safety and Antitumour Activity of ODM-201 (BAY-1841788) in Castration-resistant, CYP17 Inhibitor-naive Prostate Cancer: Results from Extended Follow-up of the ARADES Trial. Eur Urol Focus. 2017 Dec;3(6):606-614. doi: 10.1016/j.euf.2017.01.010. Epub 2017 Feb 27. PMID 28753849
- [Derived] Fizazi K, Massard C, Bono P, Jones R, Kataja V, James N, Garcia JA, Protheroe A, Tammela TL, Elliott T, Mattila L, Aspegren J, Vuorela A, Langmuir P, Mustonen M; ARADES study group. Activity and safety of ODM-201 in patients with progressive metastatic castration-resistant prostate cancer (ARADES): an open-label phase 1 dose-escalation and randomised phase 2 dose expansion trial. Lancet Oncol. 2014 Aug;15(9):975-85. doi: 10.1016/S1470-2045(14)70240-2. Epub 2014 Jun 25. PMID 24974051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 17 hospitals in Europe and in the USA
Pre-assignment Details: Patients with response or stable disease at week 12 in ARADES 3104001 study as judged by the investigator, were allowed to continue in the ARADES-EXT 3104002 extension study.
Groups:
- Patients From Arades 3104001 Dose Escalation: 200 mg/day, 400 mg/day, 600 mg/day, 1000 mg/day, 1400 mg/day, 1800 mg/day
- Patients From Arades 3104001 Dose Expansion (200mg/Day); Patients From Arades 3104001 Dose Expansion (400mg/Day); Patients From Arades 3104001 Dose Expansion (1400mg/Day): Chemotherapy-naïve and CYP17 inhibitor-naïve, Post-chemotherapy and CYP17 inhibitor-naïve, Post-CYP17 inhibitor.
Period: Overall Study
Arm/Group | Patients From Arades 3104001 Dose Escalation | Patients From Arades 3104001 Dose Expansion (200mg/Day) | Patients From Arades 3104001 Dose Expansion (400mg/Day) | Patients From Arades 3104001 Dose Expansion (1400mg/Day)
Started | 19 | 22 | 19 | 16
Completed | 19 | 22 | 19 | 16
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients From Arades 3104001 Dose Escalation | Patients From Arades 3104001 Dose Expansion (200mg/Day) | Patients From Arades 3104001 Dose Expansion (400mg/Day) | Patients From Arades 3104001 Dose Expansion (1400mg/Day) | Total
Number analyzed (Participants) | 19 | 22 | 19 | 16 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (6.1) | 66.5 (6.6) | 68.9 (8.3) | 74.6 (6.3) | 69.4 (7.3)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 19 | 22 | 19 | 16 | 76

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events from start of ODM-201 treatment (in ARADES 3104001 study) until end of study visit (in ARADES-EXT 3104002 study). Median duration on study treatment was 11,0 months.
Time Frame: From first dose of study treatment up to 4 weeks after last dose of study treatment
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Patients From Arades 3104001 Dose Escalation | Patients From Arades 3104001 Dose Expansion (200mg/Day) | Patients From Arades 3104001 Dose Expansion (400mg/Day) | Patients From Arades 3104001 Dose Expansion (1400mg/Day)
Number analyzed (Participants) | 19 | 22 | 19 | 16
participants | 19 | 22 | 19 | 16

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 4 weeks after last dose of study treatment. Median duration on study treatment was 11,0 months.
Arm/Group | Patients From Arades 3104001 Dose Escalation | Patients From Arades 3104001 Dose Expansion (200mg/Day) | Patients From Arades 3104001 Dose Expansion (400mg/Day) | Patients From Arades 3104001 Dose Expansion (1400mg/Day)
Serious Adverse Events (participants affected / at risk) | 5/19 | 7/22 | 3/19 | 4/16
Other Adverse Events (participants affected / at risk) | 19/19 | 22/22 | 19/19 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients From Arades 3104001 Dose Escalation (N=19) | Patients From Arades 3104001 Dose Expansion (200mg/Day) (N=22) | Patients From Arades 3104001 Dose Expansion (400mg/Day) (N=19) | Patients From Arades 3104001 Dose Expansion (1400mg/Day) (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Enterobacter infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 1 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Enterobacter test positive (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients From Arades 3104001 Dose Escalation (N=19) | Patients From Arades 3104001 Dose Expansion (200mg/Day) (N=22) | Patients From Arades 3104001 Dose Expansion (400mg/Day) (N=19) | Patients From Arades 3104001 Dose Expansion (1400mg/Day) (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abnormal faeces (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 3 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 9 | 0 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 3
Flatulence (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 2 | 3 | 3
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 2
Asthenia (General disorders) | 5 | 1 | 2 | 0
Chest pain (General disorders) | 1 | 0 | 2 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 5 | 3 | 5 | 8
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 3 | 2 | 1 | 5
Pain (General disorders) | 4 | 7 | 1 | 3
Peripheral swelling (General disorders) | 1 | 2 | 0 | 1
Pyrexia (General disorders) | 0 | 2 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 2 | 1 | 1
Onychomycosis (Infections and infestations) | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 1 | 0
Viral infection (Infections and infestations) | 1 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 2
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 2 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 1 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram PR prolongation (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 1
Heart rate increased (Investigations) | 0 | 1 | 0 | 0
Liver palpable (Investigations) | 0 | 0 | 1 | 0
Urine output increased (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 5 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 7 | 3 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4 | 5 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Exposed bone in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint lock (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 1 | 0
Areflexia (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 3 | 0
Headache (Nervous system disorders) | 4 | 2 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Hyporeflexia (Nervous system disorders) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 2 | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 0 | 1 | 0
Petit mal epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 3 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 3 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Bladder dilatation (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 3 | 1 | 2
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 1
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 1 | 0 | 0
Micturition frequency decreased (Renal and urinary disorders) | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 2 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary tract inflammation (Renal and urinary disorders) | 1 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 3 | 1 | 2 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 2 | 0 | 1
Penile oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Aortic arteriosclerosis (Vascular disorders) | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 1
Hot flush (Vascular disorders) | 1 | 1 | 3 | 2
Hypertension (Vascular disorders) | 2 | 2 | 2 | 3
Intermittent claudication (Vascular disorders) | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 2 | 0 | 0 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Poor peripheral circulation (Vascular disorders) | 0 | 0 | 0 | 1
Superficial vein prominence (Vascular disorders) | 1 | 0 | 0 | 0
Lymphostasis (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other